CLINICAL TRIAL: NCT05835323
Title: Initial Experience of the Treatment of Kidney Stones With the MONARCH™ Platform, Urology
Brief Title: Initial Clinical Experience With the MONARCH Platform, Urology for the Treatment of Kidney Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auris Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-URO-0001; 2021-URO-0001 (Other: Auris Health, Inc.)
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Kidney Calculi
Keywords: Nephrolithotomy, Percutaneous, Ureteroscopy, Robotic, Monarch, Kidney Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Robotic-assisted mini-Percutaneous Nephrolithotomy (PCNL) (Experimental): Participants with kidney stones will be enrolled for robotic-assisted mini-percutaneous nephrolithotomy procedure using the MONARCH Platform, Urology for removal of kidney stones. The MONARCH Platform, Urology enables electro-mechanical articulation and precise control of a flexible ureteroscope and/or a flexible mini-PCNL suction catheter for visualization and access to the urinary tract for diagnostic and therapeutic procedures.
  Interventions: Device: Robotic-assisted mini-PCNL

INTERVENTIONS:
Device: Robotic-assisted mini-PCNL — Eligible participants will be enrolled to undergo robotic-assisted PCNL using the MONARCH Platform, Urology for the removal of kidney stones. The MONARCH Platform, Urology is a novel flexible robotic device that enables the clinician to obtain both transurethral and percutaneous access to a participant's kidney under continuous visualization for therapeutic application (for example, stone removal).

SUMMARY:
The purpose of this study is to collect descriptive performance data using the MONARCH Platform, Urology (a novel robotic device) to perform mini-percutaneous nephrolithotomy (kidney stone removal) procedures. Data gathered from this study will be used to optimize the robotic platform and inform training and education material for the future users.

ELIGIBILITY:
Inclusion Criteria:

* Simple renal caliceal and/or pyelo stone(s), greater than or equal to (>=) 10 millimeter in size identified on computerized tomography (CT) scan, and appropriate for Percutaneous nephrolithotomy (PCNL) treatment according to American Urological Association (AUA) guidelines
* Normal upper tract anatomy, amenable to PCNL and ureteroscopy
* Body mass index less than (<) 40 kilogram-meter squared
* Participants with a percutaneous tract length <15 centimeter as measured by the estimation of the skin to stone or skin to appropriate calyx for treatment through a CT scan
* Participant is an appropriate candidate for a mini-PCNL based on the clinical guidelines and investigator assessment

Pre-Operative Exclusion Criteria:

* Any medical or physical condition/limitation that would contraindicate a conventional ureteroscopy or PCNL [for example, atypical interposition of visceral organs (bowel, spleen, or liver)] in the supine position. This assessment will be made by the investigator team
* Participation in any other clinical trial 30-days before and throughout the duration of the study that might impact the results
* A solitary functioning kidney
* Female subjects who are pregnant or nursing or those of childbearing potential refusing a pregnancy test
* Presence of ureteral impacted stones
* Presence of ureteral obstruction
* Presence of untreated urinary tract infection, urosepsis
* Inability to give consent
* Presence of a renal mass which has not been investigated
* Staghorn stone
* Participant has an electrically or magnetically activated implanted medical device
* Significant pharmacological anticoagulant therapy or uncorrected bleeding diathesis
* Tumor in the probable access tract area and potential malignant renal tumor

Intra-Procedure Exclusion Criteria:

- Any presenting condition discovered intra procedurally that in the opinion of the investigator would make participating in this study not in the participant's best interest. For example, participants no longer considered good candidates for a mini-PCNL procedure for the removal of the kidney stones.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Landman, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California - Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged 22 years or older with simple renal caliceal and/or pyelo stone(s), greater than or equal to 10 millimeters in size identified on computed tomography scan, and appropriate for percutaneous nephrolithotomy (PCNL) treatment according to American Urological Association guidelines were considered for the study. Participants were given the Informed Consent Form to read, ask questions, and sign prior to any study procedures being performed or data being collected.
Pre-assignment Details: This was a single-arm study where all participants received treatment with the MONARCH™ Platform, Urology system.
Units Other Than Participants: Kidney stones
Groups:
- Robotic Mini-PCNL: The MONARCH™ Platform, Urology enables electro-mechanical articulation and precise control of a flexible ureteroscope and/or a flexible mini-PCNL suction catheter for visualization and access to the urinary tract for diagnostic and therapeutic procedures.
Period: Overall Study
Arm/Group | Robotic Mini-PCNL
Started | 13; 32 Kidney stones
Completed | 13; 32 Kidney stones
Not Completed | 0; 0 Kidney stones

BASELINE CHARACTERISTICS:
Population: All 13 participants who started the study are included in all summaries of baseline characteristics, outcome measures and adverse events.
Units Other Than Participants: Kidney stones
Arm/Group | Robotic Mini-PCNL
Number analyzed (Participants) | 13
Number analyzed (Kidney stones) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Completion of the Robotic Assisted Mini-PCNL Kidney Stone Removal Procedure.
Description: Percentage of participants in whom the kidney stone treatment and removal procedure could be successfully completed with the MONARCH™ Platform, Urology.
Time Frame: Day of Procedure
Population: All 13 participants who started the study and were treated with MONARCH™ Platform, Urology.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Mini-PCNL
Number analyzed (Participants) | 13
Participants | 12

ADVERSE EVENTS:
Time Frame: 30 days post stone removal procedure
Description: An adverse event (AE) is defined as any undesirable clinical occurrence in a patient whether or not it is considered to be device related. In addition, the definition of AE applies to any event with an onset post study procedure or to any underlying diseases, present at baseline, that exacerbate in severity post study procedure. All reported AEs must be recorded in the database.
Arm/Group | Robotic Mini-PCNL
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Mini-PCNL (N=13)
Bacteraemia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Mini-PCNL (N=13)
Urinary tract infection (Infections and infestations) | 1 (1)
Ureteric injury (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a single-arm, single-center, first-in-human experience with the MONARCH™ Platform, Urology in a small set of participants without a control arm. As such the generalizability of the results obtained are limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator(s) may publish or present the Study results with prior consent of the Sponsor but will not disclose confidential information. Prior to submission by a Principal Investigator for publication or presentation, the Sponsor will be provided with the opportunity to review the submission for confidential information and accuracy.

DOCUMENTS (2):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT05835323/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT05835323/SAP_001.pdf